CLINICAL TRIAL: NCT03844490
Title: Timing of Umbilical Cord Clamping and Maternal and Neonatal Outcomes, Comparing One to Three Minutes vs. After Cessation of Cord Pulsation: a Randomized Clinical Trial
Brief Title: Timing of Umbilical Cord Clamping: One to Three Minutes vs. After Cessation of Cord Pulsation
Acronym: CORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Collaborators: Hospital Da Mulher do Recife (Unknown)
Responsible Party: Principal Investigator, Leila Katz, Coordinator of the Obstetrical Intensive Care Unit, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CORD
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Umbilical Cord
Keywords: Postpartum Hemorrhage; Neonatal jaundice; Umbilical cord
MeSH Terms: conditions — Postpartum Hemorrhage; Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Other): In this group management will be carried out as usual routine (cord clamping from one to three minutes after delivery)
  Interventions: Other: CONTROL
- CESSATION OF CORD PULSE (Experimental): In this group the umbilical cord will remain unclamped until the spontaneous pulsation stops.
  At this time, cord clamping will be made.
  Interventions: Other: CESSATION OF CORD PULSE

INTERVENTIONS:
Other: CESSATION OF CORD PULSE — In this group the umbilical cord will remain unclamped until the spontanous pulsation stops.
  At this time, cord clamping will be made.
  Arms: CESSATION OF CORD PULSE
Other: CONTROL — In this group management will be carried out as usual routine (cord clamping from one to three minutes after delivey)
  Arms: CONTROL

SUMMARY:
The timing of umbilical cord clamping has been widely discussed in the scientific community.

As part of the worldwide strategies to reduce childhood iron deficiency anemia, the incorporation of late clamping (at least one minute after delivery), has been adopted as an effective and low-cost measure for health services.

The optimal timing for clamping, ( if until 3 minutes of delivery, or later, when the cord stops spontaneous pulse), still remains controversial.

Also, doubts remain about the effect of late clamping of the umbilical cord on maternal outcomes.

This study has the hypothesis that waiting for the cessation of the cord pulsation will not bring harm to the newborn or the mother.

DETAILED DESCRIPTION:
Due to several studies showing the advantages of late clamping of the umbilical cord for the newborn child. Delayed clamping from one, up to three minutes has been associated with better adaptation of the neonate to extrauterine life, with increased supply of oxygen, iron reserve in childhood, and benefits in the neuropsychic and motor development of children. It is considered a safe technique, recommended and has been recommended by obstetrics and neonatologists throughout the world, although the exact moment for its accomplishment is not aligned between countries.

Early clamping was one of the strategies of active management in the third period of delivery in order to prevent postpartum hemorrahge (PPH), which is considered a major cause of maternal mortality worldwide. Studies have not confirmed this initial hypothesis and the balancing between the advantages for the newborn, and no evidence of advantage fot he mother has shifted the management to late cord clamping, which for most professionals consists of clamping the cord from one to three minutes after birth.

On the other hand, there are still questions regarding the possibility of prolonging the cord clamping time, for an even longer time, or even stopping the cord's pulsations, as a way to favor placental drainage, reduce the time of placental detachment and consequently decrease bleeding events. It is believed that delayed clamping after pulsations cease may contribute to the increase in the blood volume transferred to the neonate, thus increasing its iron stores without any additional harm to the health of the woman and the newborn.

The subject is new, in order to verify the impact on the occurrence of neonatal jaundice and the blood loss when the cord is clamped after the pulsations cease, since there is no detailed report in any other study on this practice. Thus, it can contribute to the available evidence on the subject, and can be included in a systematic review and enable the elucidation of questions that still need to be clarified.

The study is relevant, since the conclusions may be of great use for clinical conduct, since it is a non-invasive and cost-free method that can contribute to reduce the occurrence of iron deficiency anemia in early childhood and postpartum haemorrhage.

General objective To determine the effects of late clamping of the umbilical cord with one to three minutes vs. after pulsations on maternal and neonatal outcomes ceased.

Specific objectives

In neonates and women undergoing delayed clamping with one to three minutes and after ceasing the cord pulsations, compare:

Primary Outcomes Rate of neonatal hyperbilirubinemia, requiring phototherapy is equivalent in both groups.

Neonatal hemoglobin between 24-48 hours postpartum is higher in the intervention group.

Secondary Outcomes Neonatal Weight at birth; Apgar score in the first minute and fifth minute; Skin-to-skin contact in the first hour of life; Duration of skin-to-skin contact; Breastfeeding in the first hour; Breastfeeding until discharge; Concentration of Ht at birth and between 24-48 hours after birth; Need for admission to neonatal neonatal intensive care unit (ICU); Hyperbilirubinemia requiring exchange transfusion; Neonatal polycythemia. Maternal Postpartum blood loss; PPH (blood loss> 1,000ml); Hemoglobin (HG) and (Hematocrit) Ht levels in 24 hours postpartum; Hemoglobin levels lower than 8 g / dl in 24 hours postpartum; Time of detention less than 30 minutes; Uterine manual cleaning, uterine curettage, and manual removal of the placenta; Treatment for PPH in the first hour up to 24 hours postpartum; Hemotransfusion after delivery; Maternal death; Level of maternal satisfaction. Study design=> open randomized clinical trial The study will be conducted in Instituto de Saude Integral Prof Fernando Figueira (IMIP) and Hospital da Mulher do Recife (HMR). Sample will be composed of normal risk women, live fetus at term, hospitalized in labor and by their newborns attended during the study period in the hospitals involved in the research.

Sample size calculation The sample was calculated using the online public domain calculator, Sealed Envelope 2012, considering data from a study in which 4.36% of newborns submitted to umbilical cord clamping at three minutes presented hyperbilirubinemia requiring phototherapy, with the maximum tolerable frequency of 5.36%, to show that there is no superiority between the two ducts, with a power (1-error beta) of 90% and a level of bilateral significance of (1-alpha error) of 95% 526 patients were needed, a number that was increased to 580 patients, 290 in each group, and possible losses were predicted.

After consenting to participate a blood sample will be collected from the pregnant woman by the laboratory professional, at the obstetric screening or at the PP, immediately before delivery, and sent to the laboratory for analysis of hemoglobin and hematocrit levels. All participants will be assisted in labor and delivery performed according to the routine of the service. Only after birth, if the newborn meets the eligibility criteria, will the allocation be made to one of the two previously randomized groups, with opening of the sealed envelopes.

Data collection will be performed by the assistant researchers and professionals on duty (nurse obstetrician, obstetrician and / or nursing residents) during the daytime and night shift on weekends and holidays, filling in the 24 hours of the shift. Within 24 hours of delivery, a new blood sample from the puerperium will be collected by the laboratory employee to evaluate hemoglobin and hematocrit levels; and the newborn for evaluation of hemoglobin, hematocrit and total bilirubin levels.

Data processing and analysis The analysis of the data will be performed by a blind statistic collaborator of the test, using the statistical program Epi-Info 3.5.4. The analysis will be done by intention to treat the data and performed with the groups identified as A or B. Only at the end of the analysis, already prepared the tables, is that you will know about which group will correspond each letter.

To evaluate the association between the independent variable or predictor (clamping of the umbilical cord with one to three minutes vs. clamping after the pulsations cease) and the dependent variables (outcomes) will be constructed double-entry tables. For the primary outcome, we will work with the equivalence hypothesis and for the secondary outcomes with the hypothesis of superiority.

For the continuous numerical variables of normal distribution, Student's t-test will be used, if the normality of the distribution is not verified (Kolmogorov-Smirnov test), the Mann-Whitney test will be used. For categorical variables, the Chi-square test of association (Pearson) and Fisher's exact test, when applicable, will be used. All adopted p values will be counted. The Risk Ratio (RR) will be calculated as a measure of the relative risk, as well as the 95% Confidence Interval (95% CI). The default value of 1.0 will be assigned to the reference category.

ELIGIBILITY:
Inclusion Criteria:

(pregnant women)

* Low risk pregnancy;
* Full-term pregnancy (37 to 42 weeks);
* Single fetus;
* Cephalic presentation;
* Normal birth;
* Euthocic delivery. (newborns)
* Live birth;
* Apgar> 7 in the first minute and fifth minutes.

Exclusion Criteria:

Early clamping for any reason (indicated by assistant);

* Instrumental delivery (forceps);
* Chorioamnionitis;
* Placental abruption;
* Prolapse of umbilical cord;
* Congenital anomaly;
* Labor analgesia.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Neonatal Hyperbilirubinemia requiring phototherapy | 24 to 7 days after birth
  clinical situation where hyperbilirubinemia indicates phototherapy. The need for phototherapy will be identified from the analysis of the laboratory results of total bilirubin, applying the values established by the American Academy of Pediatrics (AAP).
Neonatal hemoglobin concentration 24-48 h postpartum | 24 to 48 hours after birth
  expressed the concentration of neonatal hemoglobin, collected between 24 and 48 hours postpartum

SECONDARY OUTCOMES:
Weight of the newborn | 1 hour postpartum
  corresponds to the measurement of the weight of the newborn, measured in grams, performed in the first hour after
Apgar Score in the first and fifth minutes | 5 minutes
  corresponds to a scale that aims to evaluate the vitality of the neonate immediately after birth in the first and fifth minutes
Skin-to-skin contact | 5 hours
  is defined as the skin-to-skin contact of the newborn with its mother immediately after delivery by placing it on the mother's chest or abdomen.
Duration of skin-to-skin contact | 5 hours
  duration of time of skin-to-skin contact of the newborn to its mother
Breastfeeding in the first hour after birth | 1 hour
  occurrence of breastfeeding in the first hour after birth
Breastfeeding until discharge | 15 days
  the occurrence of breastfeeding on a regular basis until hospital discharge
Hematocrit concentration 24-48 hours | 24-48 hours
  concentration of neonatal hematocrit from the collection of a peripheral blood sample of the newborn through the median or medial basilar vein in the left or right arm of the left or right arm between 24 and 48 hours postpartum
Need of ICU or NICU | 28 days
  the need for hospitalization of the newborn in the Intermediate Care Unit (ICU) or neonatal intensive care unit (NICU)
Hyperbilirubinemia requiring exchange transfusion | 7 days
  The need for exchange transfusion will be identified from the analysis of laboratory results of total bilirubin, applying the values established by the American Academy of Pediatrics (AAP).
Blood loss at birth | 3 hours
  amount of blood volume lost at delivery until delivery of the placenta.
Postpartum haemorrhage | 24 hours
  PPH greater than or equal to 1,000 ml of blood or blood loss accompanied by signs and symptoms of hypovolemia at 24 hours postpartum
maternal hemoglobin 24 hours postpartum | 24 hour
  indicates the amount of maternal hemoglobin 24 hours postpartum
HG < 8 g / dL | 24 hours
  maternal hemoglobin less than 8 g / dL within 24 hours of delivery
Third period duration | 3 hours
  corresponds to the time of the delivery of the placenta (started after the fetal detachment), expressed in minutes
Uterine curage | 3 hours
  need manual curage of the uterine cavity
Uterine curettage | 3 hours
  need of uterine curettage
Manual removal of the placenta | 3 hours
  need of manual removal of the placenta
Treatment of PPH | 24 hours
  need for treatment for postpartum haemorrhage in the first hour and / or up to 24 hours postpartum
Blood transfusion | 24 hours
  need of transfusion of blood products
Maternal death | 42 days
  maternal death secondary to PPH
Maternal satisfaction | 24 hours
  maternal satisfaction with the management of umbilical cord clamping with one to three minutes and after pulsations ceased. Categorical categorical variable, which can vary between very satisfied, satisfied, not satisfied, dissatisfied and very dissatisfied, according to the scale of faces.
  The satisfaction scale will be an association between the face scale (Figure 2) and the numerical scale. Each level will be clearly explained to the patient as follows:
  * 0 - Very satisfied;
  * 1 - Satisfied;
  * 2 - Unsatisfied;
  * 3 - Unsatisfied;
  * 4 - Very dissatisfied.
  For the purposes of analysis, the satisfaction will be recoded in satisfied (yes or no), corresponding yes to categories 0 and 1 above characterized.

CONTACTS AND LOCATIONS:
Overall Officials: LEILA KATZ, MD, PhD, Study Director — IMIP
Locations (1):
- Instituto Materno Infantil Prof. Fernando Figueira, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.